CLINICAL TRIAL: NCT05555238
Title: An Observational Study to Evaluate the Safety and Effectiveness of Newvast Tab(Atorvastatin) in Korean Dyslipidemia Patients
Brief Title: An Observational Study to Evaluate the Treatment of Newvast® Tab(Atorvastatin) in Korean Patients With Dyslipidemia
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-NEW-OS-1901
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-08

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; Atorvastatin; Statin
MeSH Terms: conditions — Dyslipidemias | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: single arm, single group(No interventional) — (Newvast® Tab, 10 to 80 mg daily administered per the locally approved product information)
  Other Names: Observational

SUMMARY:
In this study, dyslipidemia patients visited the institutions during the study period and the effectiveness and safety of the treatment of Newvast® Tab(Atorvastatin) in real-practice.

During the routine medical visit, according to the investigator's judgment, with diagnosis that the Newvast® Tab(Atorvastatin) prescription is appropriate, regardless of medical history and concomitant-medication, and after deciding to start treatment, patients with Dyslipidemia who agreed to participate in the study were administered Newvast® Tab(Atorvastatin).

As this study is a non-interventional observational study, all subjects received prescriptions according to the routine treatment procedure, and there were no visits or procedures required according to the observational study protocol.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, non-interventional, observational study of patients administering Atorvastatin(Newvast® Tab) to treat Dyslipidemia.

Data will be collected from patients receiving routine treatment at hospitals in South Korea. Each subject visits the institution according to the protocol that designed the follow-up visits for six months to examine the effectiveness and safety of Atorvastatin(Newvast® Tab).

This study will approved by the institutions' IRBs and is in compliance with clinical research ethics regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was diagnosed with Dyslipidemia
2. Those who voluntarily consented in writing to this study

Exclusion Criteria:

(1) Patients for whom use of Newvast® Tab is prohibited

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dyslipidemia
Sampling Method: Non-Probability Sample
Enrollment: 1716 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
The incidence of myalgia | 6 months
  The incidence of myalgia associated with Newvast® Tab(Atorvastatin) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ji-yeon Hong, PM, Study Director — Hanmi Pharmaceutical Company Limited
Locations (1):
- Hanmi Pharmaceutical Company Limited, Seoul, South Korea